CLINICAL TRIAL: NCT02972242
Title: Focused Field of View Calcium Scoring Prior to Coronary CT Angiography
Acronym: FOCUS-CCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hampton Crimm, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 396906
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Radiation Safety; Coronary Computed Tomography Angiography; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Field of View (Active Comparator): In patients randomized to undergo the modified non-contrast CT scan to assess coronary calcification burden, this study will be performed by a radiologist and cardiologist as follows: axial acquisition obtained at 70% of the R-R interval using the following parameters: rotation time 0.35 sec; collimation of 64 x 0.625mm; detector coverage of 20.0 mm; axial thickness 2.5; tube voltage 80kV and tube current 250mA. The scan length will be from 1 cm below the carina to the level beneath the proximal coronary vessels defined as the greatest diameter of the apex of the right atrium.
  Interventions: Radiation: Field of View
- Standard Field of View (Placebo Comparator): In patients randomized to standard coronary artery calcium scoring, this scan will be performed in usual axial fashion obtained at 70% of the R-R interval using the following parameters: rotation time 0.35 sec; collimation of 64 x 0.625mm; detector coverage of 20.0 mm; axial thickness 2.5; tube voltage, 120 kV and tube current 250mA. The scan length, in accordance with current protocol, will be from 1 cm below the carina through the diaphragms.
  Interventions: Radiation: Field of View

INTERVENTIONS:
Radiation: Field of View — Non-Contrast CT Scan for coronary calcium assessment prior to CT coronary angiography

SUMMARY:
Coronary computed tomography angiography (CCTA) is a frequently performed test for the diagnosis and/or exclusion of coronary artery disease (CAD) in appropriately selected patients. The performance of non-contrast computed tomography for the detection and quantification of coronary calcification is typically performed prior to CCTA in an effort to identify significant calcification which may influence subsequent data acquisition during the CCTA. However, performance of calcium scoring adds significant radiation and most coronary calcification is proximal in its location, potentially visualized using a focused non-contrast scan.

The purpose of this study is to prospectively compare the usefulness of a modified non-contrast CT, using a significantly shorter scan length and lower radiation parameters, as compared to standard coronary artery calcium scanning for the detection of coronary calcification that may influence subsequent CCTA performance.

DETAILED DESCRIPTION:
Prior to undergoing CCTA, non-contrast CT scanning of the entire heart is usually performed in adults over 50-years of age in order to assess for the presence and severity of coronary artery calcium. By providing a modified CT scan with a reduced length the same data can be obtained by the imager to ensure a high quality scan while decreasing the patient's overall radiation exposure. Our objectives and specific aims to validate our hypothesis include:

* To assess the impact on CCTA image quality using modified calcium score approach
* To determine the rate of changes in the coronary CT angiography acquisition parameters after evaluation of the modified versus standard calcium scoring scout series. Significant changes in CCTA acquisition include any of the following as compared to recommended CCTA parameters prior to scout CT performance: a change (increase or decrease) in tube current (mA) by 50, any change in tube potential (kV), change to/from retrospectively-gated CCTA, any change in padding (acquisition window), or changing to/from a high definition CT scan acquisition.
* To assess the difference in patient estimated effective radiation exposure (mSv) between the modified versus standard calcium scoring techniques.
* To assess the difference in patient estimated effective radiation exposure (mSv) of the entire CCTA study (plus calcium scoring) between groups.

Study Design Prospective, randomized single-center cohort study.

Anticipated Requirements

1. Facilities: Walter Reed National Military Medical Center

   1. Cardiology Clinic
   2. Cardiovascular Health and Interventional Radiology, Angiography and Recovery [CVHIR]
   3. Radiology Department (CT Section)
2. Duration of enrollment: 12 months
3. Budget: no additional budget is needed.

Subject Population

1. One hundred seventy-five (175) male and female adult subjects (military health beneficiaries age greater than 50 years) who are clinically referred for CCTA will be eligible for participation.
2. The Walter Reed National Military Medical Center Cardiology Department and Radiology Departments perform multiple clinically appropriate and indicated coronary CTA studies weekly (approximately 8-12), which will allow for ease of subject recruitment. Although there are other open studies using CCTA in our department there is not a lot of overlap in their requirements and should not prohibit enrollment in our study. This study will enroll both men and women of all ethnic origins aged ≥ 50 years. All subjects will consent for themselves. All patients' participation in this research and subsequent contribution to our medical knowledge notwithstanding, no intent to benefit patients from enrollment is implied or offered. Pregnant women will be excluded from enrollment based on:

   1. Verbal admission of pregnant status; OR
   2. Positive urine pregnancy test performed within 7 days of CCTA in subjects not previously known to be pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adult patients ≥ 50 years of age;
2. Suspected but without known prior history of CAD. Prior CAD is defined as a history of myocardial infarction, coronary revascularization or ≥ 50% coronary lumen stenosis on prior coronary angiography
3. Scheduled for non-emergent clinically indicated coronary CT angiography

Exclusion Criteria:

1. Prior coronary bypass graft (CABG) surgery
2. Suspicion of acute coronary syndrome (MI or unstable angina)
3. Known complex congenital heart disease
4. Evidence of ongoing or active clinical instability, including chest pain (sudden onset); cardiogenic shock; unstable blood pressure with systolic blood pressure < 90 mmHg; and severe congestive heart failure (NYHA class III or IV); or acute pulmonary embolism
5. Atrial fibrillation
6. Abnormal renal function (GFR < 60 ml/min; Creatinine > 1.5 mg/dL)
7. Concomitant participation in another clinical trial in which patient is subject to investigation drug or device
8. Pregnancy or unknown pregnancy status
9. Allergy to iodinated contrast agent
10. Contraindications to nitroglycerin
11. Unwilling or unable to give consent
12. Inability to comply with study procedures
13. Prior coronary artery calcium score and/or coronary CT angiogram

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hampton A Crimm, MD, Principal Investigator — WRNMMC Cardiology Department

REFERENCES:
- [Derived] Crimm HA, Fergestrom NM, Dye C, Philip C, Nguyen BT, Villines TC. Focused, low tube potential, coronary calcium assessment prior to coronary CT angiography: A prospective, randomized clinical trial. J Cardiovasc Comput Tomogr. 2021 May-Jun;15(3):240-245. doi: 10.1016/j.jcct.2020.08.011. Epub 2020 Aug 22. PMID 32868247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Field of View | Standard Field of View
Started | 82 | 93
Completed | 81 | 93
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 82 patients were enrolled to the Modified group. As previously mentioned, one withdrew consent immediately after randomization (i.e. prior to undergoing scan). Two additional scans within the modified group were unavailable to the PI at the time of data analysis (i.e. years after the scan, due to data migration failure)
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Field of View | Standard Field of View | Total
Number analyzed (Participants) | 79 | 93 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (5.8) | 59 (7.3) | 58 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 46 | 83
  Male | 42 | 47 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 31 | 57
  White | 37 | 50 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 2 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 93 | 172

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Quality Comparison
Description: The measurement of quality in comparison of the modified versus non-modified CCTA using a qualitative (four point scale).
  1. = Nondiagnostic: Impaired image quality that precluded appropriate evaluation of the coronary arteries due to severe motion artifacts, extensive blooming artifact, severe image noise, or insufficient contrast.
  2. = Adequate: Reduced image quality because of artifacts due to motion, image noise or low contrast attenuation, but sufficient to rule-out significant stenosis.
  3. = Good: Presence of artifacts caused by motion, image noise, coronary calcifications or low contrast, but fully preserved ability to assess the presence of luminal stenosis as well as the presence of calcified and non-calcified coronary atherosclerotic plaque.
  4. = Excellent: Complete absence of motion artifacts, strong attenuation of vessel lumen and clear delineation of vessel walls, with the ability to assess stenosis and plaque characteristics.
Time Frame: Following completion of data acquisition (i.e. CT scans) for all patients (last patient scan was 2/26/18), each outcome measure was then assessed (this process spanned approximately 3 months from March to June 2018).
Population: Within the modified group: 1 patient had previously withdrawn consent and 2 additional scans were subsequently unavailable for review at the time of measurement of the outcomes.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
score on a scale | 4 [3 to 4] | 4 [3 to 4]

2. Primary Outcome: Quantitative Quality Comparison
Description: The measurement of quality in comparison of the modified versus non-modified CCTA using a quantitative score (CCTA signal, noise, signal to noise ratio):
  image signal and noise obtained during scan analysis by placing a circular region of interest (1 cm in diameter) within the proximal ascending aorta and there measuring Hounsfield Units (HU) which is the CCTA "signal" and standard deviation of the HU within that same region (which is the "noise"), the ratio of these signal/noise is also captured by this method.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
ratio | 16.8 (6.1) | 17.9 (6.8)

3. Secondary Outcome: Number of Patients With Coronary CT Parameter Changes (mA by 50).
Description: Any changes in the cardiac CT after evaluation of the modified or standard calcium scoring in a change in milliamps by 50.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
Participants | 35 | 49

4. Secondary Outcome: Number of Patients With Coronary CT Parameter Changes (Tube Potential).
Description: Any changes in the cardiac CT after evaluation of the modified or standard calcium scoring (i.e. increasing or decreasing the tube potential)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
Participants | 23 | 22

5. Secondary Outcome: Number of Patients With Coronary CT Using High Definition Scanning.
Description: Any use of of the "high definition" scanning parameter after evaluation of the calcium burden by modified or standard calcium scoring.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
Participants | 7 | 10

6. Secondary Outcome: Number of Patients With Coronary CT Parameter Changes (Padding in Milliseconds).
Description: Any changes in the cardiac CT after evaluation of the modified or standard calcium scoring in any changes in padding (milliseconds).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
Participants | 16 | 15

7. Secondary Outcome: Comparison Radiation Exposure in Non-Con CT (Dose Length Product)
Description: The measurement of radiation exposure as DLP (measured in mSv/mGycm) in comparison of the modified versus standard calcium scoring.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mSv/mGycm
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
mSv/mGycm | 10 (6) | 53 (29)

8. Secondary Outcome: Comparison Radiation Exposure Contrast Coronary CT (Dose Length Product / Milli-sieverts)
Description: The measurement of radiation exposure difference measured as DLP/milli-sieverts of the entire CCTA study on the modified versus standard calcium scoring.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mSv/mGycm
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
mSv/mGycm | 240 (137) | 295 (190)

9. Secondary Outcome: Number of Participants for Which There Was a Scan Termination Event
Description: Number of patients whose coronary CTA scan was canceled by the imaging provider due to extreme levels of calcium noted during the modified or standard calcium scoring scan.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Field of View | Standard Field of View
Number analyzed (Participants) | 79 | 93
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Modified Field of View | Standard Field of View
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/93
Other Adverse Events (participants affected / at risk) | 0/82 | 0/93

LIMITATIONS AND CAVEATS:
single center design and relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02972242/Prot_SAP_000.pdf